CLINICAL TRIAL: NCT00723021
Title: A Phase 2a, Randomised, Double-Blind (3rd Party Open), Double-Dummy, Placebo And Active Controlled 5-Way Crossover Study To Assess The Bronchodilatory Action, Safety, Toleration And Pharmacokinetics Of Single Oral Doses Of PF-04191834 In Asthmatic Patients.
Brief Title: PF-04191834 Single Dose Bronchodilatory Study In Asthma.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B0041002
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Results first posted 2013-02-01 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2012-12

CONDITIONS: Asthma
Keywords: Bronchodilator
MeSH Terms: conditions — Asthma | interventions — zileuton

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- PF-04191834 30mg (Experimental)
  Interventions: Drug: PF-04191834
- PF-04191834 100mg (Experimental)
  Interventions: Drug: PF-04191834
- PF-04191834 2000mg (Experimental)
  Interventions: Drug: PF-04191834
- zileuton (Active Comparator)
  Interventions: Drug: zileuton
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04191834 — 30mg PF-04191834, single dose, oral dispersion + 2 x placebo tablets.
  Arms: PF-04191834 30mg
Drug: PF-04191834 — 100mg PF-04191834, single dose, oral dispersion + 2 x placebo tablets, single dose.
  Arms: PF-04191834 100mg
Drug: PF-04191834 — 2000mg PF-04191834, single dose, oral dispersion + 2 x placebo tables, single dose
  Arms: PF-04191834 2000mg
Drug: zileuton — 1200mg, 2 x 600mg tablets, single dose + placebo oral dispersion, single dose.
  Arms: zileuton
Drug: Placebo — 2 x placebo tablets + placebo oral dispersion, single dose.
  Arms: placebo

SUMMARY:
Study to determine the bronchodilatory effects of PF-04191834 compared with zileuton in patients with asthma

ELIGIBILITY:
Inclusion Criteria:

* Persistent mild/moderate asthma for at least 6 months.
* Reduced lung function
* Reversible airway obstruction

Exclusion Criteria:

* Pregnant/nursing females.
* Liver function tests greater than upper limit of normal (ULN)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2008-07; Primary Completion 2008-12 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, North Dartmouth, Massachusetts
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Omaha, Nebraska

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0041002&StudyName=PF-04191834%20Single%20Dose%20Bronchodilatory%20Study%20In%20Asthma.

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Sequence 1: Placebo/Zileuton CR 1200 mg/PF-04191834 30 mg/PF-04191834 2000 mg/PF-04191834 100 mg
- Treatment Sequence 2: PF-04191834 100 mg/PF-04191834 30 mg/PF-04191834 2000 mg/Placebo/Zileuton CR 1200 mg
- Treatment Sequence 3: PF-04191834 2000 mg/PF-04191834 100 mg/Zileuton CR 1200 mg/PF-04191834 30 mg/Placebo
- Treatment Sequence 4: PF-04191834 30 mg/Placebo/PF-04191834 100 mg/Zileuton CR 1200 mg/PF-04191834 2000 mg
- Treatment Sequence 5: Zileuton CR 1200 mg/PF-04191834 2000 mg/Placebo/PF-04191834 100 mg/PF-04191834 30 mg
Period: Intervention Period 1
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4 | Treatment Sequence 5
Started | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Intervention Period 2
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4 | Treatment Sequence 5
Started | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Intervention Period 3
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4 | Treatment Sequence 5
Started | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Intervention Period 4
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4 | Treatment Sequence 5
Started | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Period: Intervention Period 5
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4 | Treatment Sequence 5
Started | 3 | 3 | 3 | 3 | 2
Completed | 3 | 3 | 3 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants receiving any of the 5 treatments (PF-04191834 30 mg, PF-04191834 100 mg, PF-04191834 2000 mg, Zileuton CR 1200 mg and Placebo) in a randomized fashion first
Arm/Group | All Participants
Number analyzed (Participants) | 15
Age Continuous [Mean (Standard Deviation); unit: years] | 33.5 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Race/Ethnicity, Customized [Number; unit: participants]
  White | 12
  Black | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1)
Description: The FEV1 is the maximal volume of air that can be forcefully exhaled in one second
Time Frame: Baseline, 12 hours (hrs) post-dose
Population: All enrolled participants treated who had at least 1 concentration in at least 1 treatment period
Measure: Mean (Standard Deviation); unit: L
Groups:
- Placebo: Participants received a single oral dose of placebo for zileuton CR tablets or placebo for PF-04191834 oral aqueous dispersion in any treatment period
- PF-04191834 30 mg: Participants received a single oral dose of PF-04191834 30 mg in any treatment period
- PF-04191834 100 mg: Participants received a single oral dose of PF-04191834 100 mg single dose in any treatment period
- PF-04191834 2000 mg: Participants received a single oral dose of PF-04191834 2000 mg in any treatment period
- Zileuton CR 1200 mg: Paticipants received a single oral dose of zileuton CR 1200 mg (2 x 600 mg tablets) in any treatment period
Arm/Group | Placebo | PF-04191834 30 mg | PF-04191834 100 mg | PF-04191834 2000 mg | Zileuton CR 1200 mg
Number analyzed (Participants) | 15 | 14 | 15 | 15 | 15
L
  Baseline | 2.624 (0.3939) | 2.626 (0.3860) | 2.585 (0.5200) | 2.579 (0.4131) | 2.609 (0.4502)
  Change at 12 Hours Postdose | 0.064 (0.3098) | 0.164 (0.1859) | 0.152 (0.2072) | 0.265 (0.3047) | 0.131 (0.1566)

2. Primary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1)
Description: The FEV1 is the maximal volume of air that can be forcefully exhaled in one second
Time Frame: Baseline, 24 hours (hrs) post-dose
Population: All enrolled participants treated who had at least 1 concentration in at least 1 treatment period
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Placebo | PF-04191834 30 mg | PF-04191834 100 mg | PF-04191834 2000 mg | Zileuton CR 1200 mg
Number analyzed (Participants) | 15 | 14 | 15 | 15 | 15
L
  Baseline | 2.624 (0.3939) | 2.626 (0.3860) | 2.585 (0.5200) | 2.579 (0.4131) | 2.609 (0.4502)
  Change at 24 Hours Postdose | 0.122 (0.2553) | 0.014 (0.2318) | 0.103 (0.2616) | 0.162 (0.1559) | 0.151 (0.1338)

3. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC)
Description: The FVC is the maximal volume of air that can be exhaled from full inhalation by exhaling as forcefully and rapidly as possible
Time Frame: Baseline, 12 hours (hrs) post-dose
Population: All enrolled participants treated who had at least 1 concentration in at least 1 treatment period
Measure: Mean (Standard Deviation); unit: L
Groups:
- Placebo: Each subject received 2 x placebo tablets ( for zileuton 600 mg tablets) + placebo oral dispersion (for PF-04191834), single dose
- PF-04191834 30 mg: Each subject received PF-04191834 30 mg, single dose, oral dispersion + 2 x placebo tablets
- PF-04191834 100 mg: Each subject received PF-04191834 100 mg, single dose, oral disersion + 2 x placebo tablets, single dose
- Zileuton CR 1200 mg: Each subject received zileuton CR 1200 mg, 2x600 mg tablets, single dose + placebo oral dispersion, single dose
Arm/Group | Placebo | PF-04191834 30 mg | PF-04191834 100 mg | PF-04191834 2000 mg | Zileuton CR 1200 mg
Number analyzed (Participants) | 15 | 14 | 15 | 15 | 15
L
  Baseline | 3.852 (0.8865) | 3.891 (0.8625) | 3.720 (0.8930) | 3.792 (0.9100) | 3.821 (0.9914)
  Change at 12 Hours Postdose | 0.025 (0.3306) | 0.284 (0.4150) | 0.210 (0.4792) | 0.266 (0.3184) | 0.140 (0.2750)

4. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC)
Description: as for outcome 3
Time Frame: Baseline,24 hours (hrs) post-dose
Population: All enrolled participants treated who had at least 1 concentration in at least 1 treatment period
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Placebo | PF-04191834 30 mg | PF-04191834 100 mg | PF-04191834 2000 mg | Zileuton CR 1200 mg
Number analyzed (Participants) | 15 | 14 | 15 | 15 | 15
L
  Baseline | 3.852 (0.8865) | 3.891 (0.8625) | 3.720 (0.8930) | 3.792 (0.9100) | 3.821 (0.9914)
  Change at 24 Hours Postdose | 0.162 (0.2322) | 0.051 (0.2839) | 0.229 (0.3657) | 0.171 (0.2070) | 0.219 (0.2977)

5. Secondary Outcome: Change From Baseline in Forced Expiratory Flow Between 25 and 75% of Vital Capacity (FEF25-75)
Description: The FEF25-75 is the forced expiratory flow between 25 and 75% of vital capacity
Time Frame: Baseline, 12 hours (hrs) post-dose
Population: All enrolled participants treated who had at least 1 concentration in at least 1 treatment period
Measure: Mean (Standard Deviation); unit: L/Sec
Arm/Group | Placebo | PF-04191834 30 mg | PF-04191834 100 mg | PF-04191834 2000 mg | Zileuton CR 1200 mg
Number analyzed (Participants) | 15 | 14 | 15 | 15 | 15
L/Sec
  Baseline | 1.951 (0.4550) | 1.901 (0.4228) | 1.807 (0.4452) | 1.915 (0.4488) | 1.959 (0.4378)
  Change at 12 Hours Postdose | 0.091 (0.3556) | 0.340 (0.4238) | 0.269 (0.3033) | 0.297 (0.3871) | 0.187 (0.3757)

6. Secondary Outcome: Change From Baseline in Forced Expiratory Flow Between 25 and 75% of Vital Capacity (FEF25-75)
Description: The FEF25-75 is the forced expiratory flow between 25 and 75% of vital capacity
Time Frame: Baseline, 24 hours (hrs) post-dose
Population: All enrolled participants treated who had at least 1 concentration in at least 1 treatment period
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Placebo | PF-04191834 30 mg | PF-04191834 100 mg | PF-04191834 2000 mg | Zileuton CR 1200 mg
Number analyzed (Participants) | 15 | 14 | 15 | 15 | 15
L
  Baseline | 1.951 (0.4550) | 1.901 (0.4228) | 1.807 (0.4452) | 1.915 (0.4488) | 1.959 (0.4378)
  Change at 24 Hours Postdose | 0.146 (0.3049) | 0.038 (0.1952) | 0.196 (0.2169) | 0.151 (0.2030) | 0.208 (0.3483)

7. Other Pre Specified Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time Frame: Pre-dose, 2, 4, 5, 6, 10, 14 and 24 hours following dosing in each period.
Population: All enrolled subjects treated who have at least one of the PK parameters of interest in at least one treatment period.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | PF-04191834 30 mg | PF-04191834 100 mg | PF-04191834 2000 mg
Number analyzed (Participants) | 14 | 15 | 15
ng*h/mL | 1979 (482) | 5547 (1388) | 29990 (8812)

8. Other Pre Specified Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Pre-dose, 2, 4, 5, 6, 10, 14 and 24 hours following dosing in each period.
Population: All enrolled subjects treated who have at least one of the PK parameters of interest in at least one treatment period.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04191834 30 mg | PF-04191834 100 mg | PF-04191834 2000 mg
Number analyzed (Participants) | 14 | 15 | 15
ng/mL | 154 (29) | 426 (118) | 2146 (410)

9. Other Pre Specified Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: Pre-dose, 2, 4, 5, 6, 10, 14 and 24 hours following dosing in each period.
Measure: Median (Full Range); unit: hrs
Arm/Group | PF-04191834 30 mg | PF-04191834 100 mg | PF-04191834 2000 mg
Number analyzed (Participants) | 14 | 15 | 15
hrs | 6 [5 to 14] | 6 [4 to 14] | 10 [4 to 14]

10. Other Pre Specified Outcome: Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Pre-dose, 2, 4, 5, 6, 10, 14 and 24 hours following dosing in each period.
Population: Since the PK sample collection only occurred until 24 hours and the approximate t1/2 at all doses appeared to be >10 hours, t1/2 and area under the plasma concentration versus time curve until infinity (AUCinf) are not reported at any dose level.
Arm/Group | PF-04191834 30 mg | PF-04191834 100 mg | PF-04191834 2000 mg
Number analyzed (Participants) | 0 | 0 | 0

11. Other Pre Specified Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)]
Description: AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8).
Time Frame: 14 and 24 hours following dosing in each period.
Population: as for outcome 10
Arm/Group | PF-04191834 30 mg | PF-04191834 100 mg | PF-04191834 2000 mg
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Placebo: Participants received single oral dose of placebo for zileuton CR tablets or placebo for PF-04191834 oral aqueous dispersion in any treatment period
- Zileuton CR 1200 mg: Paticipants received single oral dose of zileuton CR1200 mg (2 x 600 mg tablets) in any treatment period
Arm/Group | Placebo | PF-04191834 30 mg | PF-04191834 100 mg | PF-04191834 2000 mg | Zileuton CR 1200 mg
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 9/15 | 4/14 | 10/15 | 4/15 | 12/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=15) | PF-04191834 30 mg (N=14) | PF-04191834 100 mg (N=15) | PF-04191834 2000 mg (N=15) | Zileuton CR 1200 mg (N=15)
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Viral upper respiratory tract (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 1 | 1 | 1
Headache (Nervous system disorders) | 2 | 3 | 1 | 1 | 5
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.